CLINICAL TRIAL: NCT00248911
Title: The Effect Of Meditation On Quality Of Life In Women With Breast Cancer And Other Gynecological Cancers:Avon Program for Meditation and Healing
Brief Title: The Effect Of Meditation On Quality Of Life In Women With Breast Cancer And Other Gynecological Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0209005792
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancers; Gynecologic Cancer
Keywords: Breast cancer; Gynecologic cancers; Meditation; Stress-reduction; Cognitive-affective behavioral learning
MeSH Terms: conditions — Breast Neoplasms | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness based meditation program (Experimental): Meditation and Breast Cancer: Subjects will participate in an intervention consisting of group and individual instruction in a meditation-based practice of stress-reduction and cognitive-affective-behavioral learning.
  Interventions: Behavioral: Mindfulness based meditation program

INTERVENTIONS:
Behavioral: Mindfulness based meditation program — Subjects will participate in an intervention consisting of group and individual instruction in a meditation-based practice of stress-reduction and cognitive-affective-behavioral learning.
  Other Names: Meditation and Breast Cancer

SUMMARY:
Women with breast cancer and other gynecologic cancers often suffer significant distress and disability from their disease. A practice of meditation-based stress reduction and cognitive-affective-behavioral learning may help women with these conditions decrease their suffering and improve their quality of life.

DETAILED DESCRIPTION:
The objective of this project in women recently treated for breast or other gynecologic cancer is to determine whether an intervention program consisting of group and individual instruction in a meditation-based practice of stress-reduction and cognitive-affective-behavioral learning has the potential for reducing disabling distress and improving quality of life in a population vulnerable to the progression or recurrence of disease. Quality of life will be assessed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All women with stage I-III breast or other gynecologic cancer who have received treatment within the preceding year will be eligible for inclusion in the study.

Exclusion Criteria:

* Patients who refuse to participate will be excluded
* Patients with Metastatic cancer are excluded.

Ages: 18 Years to 101 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2003-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Quality of life will be assessed by within patient differences in the FACT-G (General Functional Assessment of Cancer Treatment Scale), as well as with the disease specific subscales at baseline and at 12 months. | Subjects will complete questionnaires at baseline and closeout. Patients will participate in the meditation program weekly for 20 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University; Joseph Loizzo, MD,PhD, Principal Investigator — Center for Complementary and Intergrative Medicine, New York Presbyterian Hospital-Weill Cornell Medical College
Locations (1):
- Weill Cornell Medical College-New York Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD